CLINICAL TRIAL: NCT06551896
Title: Pemigatinib and Immune Checkpoint Inhibitor Treated FGFR1/2/3 Alteration Advanced Solid Tumor: a Single Arm, Multiple Center, Phase II Study (Pigeon Study)
Brief Title: Pemigatinib and Immune Checkpoint Inhibitor Treated FGFR1/2/3 Alteration Advanced Solid Tumor
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, qintao, associate chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-546-01
Record Dates: First submitted 2024-07-22; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Urothelial Carcinoma; Breast Neoplasms; Lung Cancer; Gastric Cancer; Soft Tissue Sarcoma; Other Carcinoma
Keywords: Pemigatinib; FGFR1/2/3 alteration; Solid tumor
MeSH Terms: conditions — Carcinoma, Transitional Cell; Breast Neoplasms; Lung Neoplasms; Stomach Neoplasms; Sarcoma; Carcinoma | interventions — pemigatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pemigatinib combined with immune checkpoint inhibitor (Experimental): Pemigatinib 13.5mg，two weeks on and one week off, and with immune checkpoint inhibitor selected by investigator.
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib and immune checkpoint inhibitors

SUMMARY:
This prospective phase Il study is aim to evaluate the efficacy and safety of FGFR inhibitor combined with immune checkpoint inhibitors in FGFR1/2/3 variant advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Histologically or cytologically confirmed unresectable advanced solid tumors with failure or intolerance to standard treatments;
* At least one measurable lesion per RECIST v1.1 criteria;
* Gene testing confirms FGFR1/2/3 variants, including but not limited to mutations, fusions/rearrangements in solid tumors;
* Patients have not previously used specific small molecule multi-target inhibitors of the FGFR pathway, as assessed by investigators, and have been treated with immune checkpoint inhibitors;
* ECOG performance status of 0-1;
* Expected survival time > 3 months;
* Laboratory criteria:

  1. Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L in the past 14 days without granulocyte colony-stimulating factor;
  2. Platelets ≥ 100 x 10⁹/L without transfusion in the past 14 days;
  3. Hemoglobin > 9 g/dL in the last 14 days without transfusion or erythropoietin;
  4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN), or total bilirubin > ULN but direct bilirubin ≤ ULN;
  5. AST, ALT ≤ 2.5 x ULN (≤ 5 x ULN in patients with liver metastasis);
  6. Serum creatinine ≤ 1.5 x ULN and creatinine clearance (Cockcroft-Gault) ≥ 50 ml/min;
  7. Good coagulation function, defined as INR or PT ≤ 1.5 x ULN. If on anticoagulant therapy, PT should be within the therapeutic range of anticoagulants;
* Female subjects of reproductive age must have a negative urine or serum pregnancy test within 3 days prior to the first dose (Cycle 1, Day 1). If the urine test is inconclusive, a blood test is required. Non-reproductive females are defined as post-menopausal for at least one year or surgically sterile;
* Subjects with reproductive potential must use contraception with an annual failure rate of less than 1% during treatment and for 120 days after the last study drug dose (or 180 days after the last chemotherapy dose).

Exclusion Criteria:

* Diagnosis of other malignancies within 3 years before the first dose, except for certain treated skin carcinomas and in-situ carcinomas;
* Previous treatment with selective FGFR inhibitors;
* Receipt of other investigational drugs within 21 days or antitumor drugs within 14 days before the first dose;
* Unresolved toxicity from prior treatments unless ≤ Grade 1 or related to alopecia or fatigue;
* Known symptomatic CNS metastasis or carcinomatous meningitis. Stable patients post-treatment with no evidence of progression may be eligible if steroid-free for at least 14 days;
* History of allogeneic organ or hematopoietic stem cell transplantation;
* Abnormal laboratory parameters:

  1. Serum phosphate > 1.5 x ULN;
  2. Elevated serum calcium or albumin-adjusted calcium outside the reference range;
* Known HIV infection or positive HIV test;
* Active or poorly controlled serious infection;
* Need for drainage treatment for pleural effusion, ascites, or pericardial effusion;
* Active hepatitis B or C infection with high viral load, or positive HBsAg or anti-HCV antibodies. Patients on antiviral therapy must meet lower thresholds;
* Significant uncontrolled heart disease, including recent MI, severe heart failure, or uncontrolled arrhythmias;
* Clinically significant ECG changes or history of significant cardiac issues; Screening QTcF interval > 480 ms, or JTc interval if applicable, must be ≤ 340 ms;
* Uncontrolled hypertension despite treatment;
* Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh grade B or higher cirrhosis;
* Major surgery within 4 weeks before the first dose or planned major surgery during the study;
* Unresolved complications from prior surgery;
* Pregnant or breastfeeding women, or those planning to become pregnant during the study period and for safety follow-up;
* Radiotherapy within 4 weeks before the first dose, except for non-CNS palliative radiotherapy with a 2-week washout period;
* History of systemic electrolyte imbalance or ectopic soft tissue calcification;
* Clinically significant corneal or retinal disease;
* Use of potent CYP3A4 inhibitors or inducers within 14 days or 5 half-lives before the first dose;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | every 8 weeks during treatment
  the proportion of patients with tumor shrinkage with CR and PR over 4 weeks.

SECONDARY OUTCOMES:
Disease control rate（DCR） | every 8 weeks during during treatment
  The proportion of patients with CR, PR and SD.
Progression-free survival （PFS） | every 8 weeks during treatment
  PFS was defined as the time from random assignment to progression or death. Patients alive who had not experienced progression as of the analysis cutoff date were censored at the last disease assessment.
Overall survival（OS） | every 8 weeks during treatment
  OS was defined as the time from random assignment to death. For patients alive at the data cutoff date, OS was censored at the last follow-up date.